CLINICAL TRIAL: NCT01769742
Title: Use of Early Mobilisation to Reduce Incidence of Hospital Acquired Pneumonia in Medical Inpatients
Brief Title: Early Mobility Bundle to Prevent Hospital Acquired Pneumonia (HAP) in Medical Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other)
Responsible Party: Principal Investigator, Alice Turner, Clinician Scientist and Honorary Consultant Physician, University of Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG-12-237
Record Dates: First submitted 2012-11-27; First posted 2013-01-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Hospital Acquired Pneumonia
Keywords: Pneumonia; promotion of activity
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobility bundle (Experimental): Delivery of early targeted physiotherapy to patients on the interventional wards; to comprise assessment and communication of mobility to ward staff and patient, provision of mobility aids, guidance and encouragement to patient and staff to allow patient to dress and mobilise independently if clinically safe to do so
  Interventions: Behavioral: Early mobility bundle
- Usual care (No Intervention): Usual physiotherapy service only

INTERVENTIONS:
Behavioral: Early mobility bundle
  Arms: Early mobility bundle

SUMMARY:
Hospital acquired pneumonia (HAP) is a common complication of extended hospital stay. In surgical specialities and critical care early physiotherapy is a recognised way of preventing such infections, and reducing length of hospital stay (LOS), however prevention of this problem is less well studied in medical inpatients.

The investigators propose a pilot study to assess the impact of introducing an early mobilisation strategy to general medical and respiratory wards at an acute Trust in the United Kingdom (UK). The investigators will recruit all new admissions to each of 2 respiratory and 2 elderly care wards - 1 of each ward type will be allocated to receive extra physiotherapy input targeting new admissions for early mobilisation. Patients' usual mobility, current mobility and actual activity levels will be studied by accelerometer and simple patient questionnaire in the first 48 hours of admission, and compared between groups. Incidence of HAP and total LOS will be recorded and compared between groups.

The investigators hypotheses are that the physiotherapy intervention will increase activity levels, reduce incidence of HAP and reduce LOS. The latter may result in cost savings to the National Health Service (NHS), which the investigators will model using local tariff data.

The investigators plan to use our data to power a larger randomised controlled study, or if the intervention is a marked success, such that a control group would be unethical, then a wider service development and evaluation programme.

ELIGIBILITY:
Inclusion Criteria:

* Any medical inpatient

Exclusion Criteria:

* Nil for main study
* Immobile patients and those unable to consent will be excluded from the sub-study using activity reporting and monitoring by Actigraph

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1178 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hospital acquired pneumonia | Duration of hospital stay (up to 12 days)
  The average length of stay is 8 days on the respiratory ward and 12 days on elderly care. This is the time period in which incidence of hospital acquired pneumonia will be measured, and expressed as incidence/week of stay. Patients whose length of stay is lower or higher than average will not be excluded.

SECONDARY OUTCOMES:
Length of hospital stay in days | Duration of hospital stay (up to 12 days)
  The average length of stay is 8 days on the respiratory ward and 12 days on elderly care. This is the time period in which incidence of hospital acquired pneumonia will be measured. Patients whose length of stay is lower or higher than average will not be excluded
Incidence of falls | Duration of hospital stay (up to 12 days)
  The average length of stay is 8 days on the respiratory ward and 12 days on elderly care. This is the time period in which incidence of hospital acquired pneumonia will be measured. Patients whose length of stay is lower or higher than average will not be excluded
Incidence of pressure area problems | Duration of hospital stay (up to 12 days)
  The average length of stay is 8 days on the respiratory ward and 12 days on elderly care. This is the time period in which incidence of hospital acquired pneumonia will be measured. Patients whose length of stay is lower or higher than average will not be excluded

OTHER OUTCOMES:
Activity levels as reported by patient | Days 1 and 2 of admission to ward
Activity levels as measured by Actigraph | Day 1 and 2 of admission to ward

CONTACTS AND LOCATIONS:
Overall Officials: Alice Turner, Principal Investigator — University of Birmingham
Locations (1):
- Heart of England NHS Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Result] Stolbrink M, McGowan L, Saman H, Nguyen T, Knightly R, Sharpe J, Reilly H, Jones S, Turner AM. The Early Mobility Bundle: a simple enhancement of therapy which may reduce incidence of hospital-acquired pneumonia and length of hospital stay. J Hosp Infect. 2014 Sep;88(1):34-9. doi: 10.1016/j.jhin.2014.05.006. Epub 2014 Jun 20. PMID 25063011